CLINICAL TRIAL: NCT05237310
Title: Dual Tandem Study Comparing the Adenoma Detection and Miss-rate of Standard Colonoscopy to That of Artificial Intelligence (CAD-EYE) and to That of Artificial Intelligence (CAD-EYE) and G-EYE® Aided Colonoscopy
Brief Title: Comparing Detection of Standard Colonoscopy, CAD-EYE and Combined CAD-EYE and G-EYE® Aided Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Smart Medical Systems Ltd. (Industry)
Collaborators: Fujifilm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: G-EYE 15076
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: G-EYE; Colonoscopy; CAD-EYE; Adenoma; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of four groups (arms), Group A1, A2, B1 and B2:
  Group A1: Subjects will undergo standard colonoscopy immediately followed by CAD-EYE colonoscopy (both procedures performed by the same endoscopist in the same sedation session). Group A2: Subjects will undergo CAD-EYE colonoscopy immediately followed by standard colonoscopy (both procedures performed by the same endoscopist in the same sedation session). Group B1: Subjects will undergo standard colonoscopy immediately followed by combined CAD-EYE and G-EYE colonoscopy (both procedures performed by the same endoscopist in the same sedation session). Group B2: Subjects will undergo combined CAD-EYE and G-EYE colonoscopy immediately followed by standard colonoscopy (both procedures performed by the same endoscopist in the same sedation session).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Colonoscopy followed by CAD-EYE (Active Comparator): Subjects will undergo standard colonoscopy immediately followed by CAD-EYE colonoscopy (both procedures performed by the same endoscopist in the same sedation session).
  Interventions: Device: Standard Colonoscopy; Device: CAD-EYE
- CAD-EYE followed by Standard Colonoscopy (Active Comparator): Subjects will undergo CAD-EYE colonoscopy immediately followed by standard colonoscopy (both procedures performed by the same endoscopist in the same sedation session).
  Interventions: Device: Standard Colonoscopy; Device: CAD-EYE
- Standard Colonoscopy followed by combined CAD-EYE and G-EYE colonoscopy (Active Comparator): Subjects will undergo standard colonoscopy immediately followed by combined CAD-EYE and G-EYE colonoscopy (both procedures performed by the same endoscopist in the same sedation session).
  Interventions: Device: Standard Colonoscopy; Device: G-EYE Colonoscopy; Device: CAD-EYE
- Combined CAD-EYE and G-EYE colonoscopy followed by Standard Colonoscopy (Active Comparator): Subjects will undergo combined CAD-EYE and G-EYE colonoscopy immediately followed by standard colonoscopy (both procedures performed by the same endoscopist in the same sedation session).
  Interventions: Device: Standard Colonoscopy; Device: G-EYE Colonoscopy; Device: CAD-EYE

INTERVENTIONS:
Device: Standard Colonoscopy — Standard Colonoscopy using a standard Fujifilm colonoscope
Device: G-EYE Colonoscopy — G-EYE Colonoscopy performed using SMART Medical G-EYE Colonoscope
  Arms: Combined CAD-EYE and G-EYE colonoscopy followed by Standard Colonoscopy; Standard Colonoscopy followed by combined CAD-EYE and G-EYE colonoscopy
Device: CAD-EYE — Colonoscopy performed using with the aid of Fujifilm CAD-EYE artificial intelligence

SUMMARY:
The purpose of this study is to compare the additional diagnostic yield over Standard Colonoscopy (i.e., the adenoma miss-rate reduction) obtained by performing CADEYE and G-EYE® aided colonoscopy, vs. the additional diagnostic yield over Standard Colonoscopy (i.e., the adenoma miss-rate reduction) obtained by performing CAD-EYE aided colonoscopy.

DETAILED DESCRIPTION:
The purpose of this study is to compare the additional diagnostic yield over Standard Colonoscopy (i.e., the adenoma miss-rate reduction) obtained by performing CADEYE and G-EYE® aided colonoscopy, vs. the additional diagnostic yield over Standard Colonoscopy (i.e., the adenoma miss-rate reduction) obtained by performing CAD-EYE aided colonoscopy. This is a single-center, four-arm dual-tandem, randomized, open-label study intended to compare the additional detection yield beyond standard colonoscopy obtained by performing combined CAD-EYE and G-EYE® high definition colonoscopy vs. the additional detection yield beyond standard colonoscopy obtained by performing CAD-EYE high definition colonoscopy. Consecutive adult subjects who were referred for elective colonoscopy will be asked to enroll into this randomized clinical study if the candidate meets the study inclusion and exclusion criteria

ELIGIBILITY:
Inclusion Criteria:

1. Screening and surveillance population for Adenoma and CRC.
2. Subjects age is at least 18 years
3. The patient must understand and sign a written informed consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of hereditary polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with prior colonic surgery (exclusion appendectomy)
6. Subjects with a history of radiation therapy to abdomen or pelvis;
7. Pregnant or lactating female subjects;
8. Subjects who are currently enrolled in another clinical investigation.
9. Subjects with current oral or parenteral use of anticoagulants, not considered eligible by the investigator.
10. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
11. Any patient condition deemed too risky for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Additional Adenoma Detection | Upon histology results (up to 30 days)
  Additional adenoma detection yield (represented by the miss rate) of CAD-EYE and G-EYE® colonoscopy over standard colonoscopy compared to the additional adenoma detection yield of CAD-EYE aided colonoscopy over standard colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator — Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH
Locations (1):
- Helios Dr. Horst Schmidt Kliniken Wiesbaden GmbH, Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: No